CLINICAL TRIAL: NCT00070135
Title: A Phase II Study Of Allogeneic Transplant For Older Patients With AML In First Morphologic Complete Remission Using A Non-Myeloablative Preparative Regimen
Brief Title: Fludarabine and Busulfan Followed by Allogeneic Stem Cell Transplant in Treating Older Patients With Acute Myeloid Leukemia in First Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-100103; CDR0000330001 (Registry Identifier: NCI Physician Data Query); NCI-2009-00438 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome
Keywords: adult acute myeloid leukemia in remission; secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities
MeSH Terms: conditions — Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Filgrastim; Antilymphocyte Serum; Busulfan; fludarabine phosphate; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (fludarabine, busulfan, allogeneic PBSC) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine IV over 30 minutes on days -7 to -3 and busulfan IV over 2 hours 4 times per day (every 6 hours) on days -4 and -3.
  GVHD PROPHYLAXIS: Patients receive tacrolimus PO or IV BID on days -2 with taper between days 90-120, and stopping by days 150-180. Patients also receive methotrexate IV on days 1, 3, 6, and 11 and rabbit antithymocyte globulin IV over 4-6 hours on days -4 through -2.
  ALLOGENEIC PBSC: Patients undergo allogeneic PBSC transplant on day 0. Patients then receive filgrastim SC daily beginning on day 12 and continuing until blood counts recover.
  Interventions: Biological: filgrastim; Biological: Anti-Thymocyte Globulin; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim — Given SC
Biological: Anti-Thymocyte Globulin — Given IV
Drug: busulfan — Given IV
Drug: fludarabine phosphate — Given IV
Drug: methotrexate — Given IV
Drug: tacrolimus — Given PO or IV
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSC transplantation
  Other Names: HSC, HSCT

SUMMARY:
This phase II trial studies how well fludarabine and busulfan followed by a donor (allogeneic) stem cell transplant work in treating older patients with acute myeloid leukemia that is in first complete remission. Giving low doses of chemotherapy, such as fludarabine and busulfan, before a donor peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stops the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving tacrolimus, methotrexate, and rabbit antithymocyte globulin before or after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if allogeneic transplantation from a matched sibling or unrelated donor using a non-myeloablative preparative regimen results in a 2-year disease-free survival (DFS) that is better than historical results using standard chemotherapy.

SECONDARY OBJECTIVES:

I. Determine 2-year actuarial risks of transplant-related mortality, acute and chronic graft-versus-host (GVHD) disease and relapse among patients with acute myeloid leukemia (AML) in first complete remission (CR1) following a non-myeloablative preparative regimen.

II. To examine recovery of T and B cell number and function following non-myeloablative stem cell transplant.

III. To examine the time course of T, B and myeloid progenitor chimerism following this preparative regimen.

IV. To characterize the pharmacokinetics of intravenous busulfan used in a non-myeloablative preparation regimen in AML patients age >= 60 years.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive fludarabine intravenously (IV) over 30 minutes on days -7 to -3 and busulfan IV over 2 hours 4 times per day (every 6 hours) on days -4 and -3.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive tacrolimus orally (PO) or IV twice daily (BID) on days -2 with taper between days 90-120, and stopping by days 150-180. Patients also receive methotrexate IV on days 1, 3, 6, and 11 and rabbit antithymocyte globulin IV over 4-6 hours on days -4 through -2.

ALLOGENEIC PERIPHERAL BLOOD STEM CELL TRASNPLANTATION (PBSC): Patients undergo allogeneic PBSC transplant on day 0. Patients then receive filgrastim subcutaneously (SC) daily beginning on day 12 and continuing until blood counts recover.

Patients are followed monthly for 1 year, every 3 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
Eligibility Criteria:

* Patients with acute myeloid leukemia (AML) (excluding French-American-British [FAB] classification system M3) who have achieved a first morphologic complete remission and who meet the criteria below; patients with preceding myelodysplastic syndrome (MDS) or treatment-related AML are eligible; patients with prior central nervous system (CNS) involvement are eligible as long as disease is in remission at transplant; patients with acute leukemia following blast transformation of prior chronic myeloid leukemia (CML) or other myeloproliferative disease are excluded
* Complete remission (CR) will be defined according to the revised recommendations of the International Working Group (24) as all of the following:

  * Normal bone marrow morphology with < 5% blasts
  * Absolute neutrophil count (ANC) > 1,000/uL, referring to the count needed to confirm that the patient achieved a CR
  * Platelet count > 100,000/uL
  * No extramedullary leukemia
  * No blasts in peripheral blood
* CR was achieved after one or two (but no more than two) cycles of induction chemotherapy with standard cytotoxic chemotherapy (e.g., cytarabine and an anthracycline) or after no more than four cycles of a hypomethylating agent containing regimen including either 5-azacytidine or decitabine
* Patients may have received as many as but no more than two cycles of consolidation therapy prior to transplant; any consolidation regimen that does not require transplant can be used; no more than 6 months can elapse from documentation of morphologic CR to transplant; the platelet count does not need to be > 100,000/uL after consolidation, as long as the bone marrow assessment prior to transplant does not show relapse
* Identification of hematopoietic cell donor
* >= 4 weeks since prior chemotherapy, radiation therapy, and surgery
* Performance status 0-2
* Diffusion capacity of carbon monoxide (DLCO) > 40% with no symptomatic pulmonary disease
* Left ventricular ejection fraction (LVEF) by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) >= 30%
* No uncontrolled diabetes mellitus or active serious infection requiring antibiotics
* No known hypersensitivity to E. coli-derived products
* No human immunodeficiency virus (HIV) infection
* Calculated creatinine clearance >= 40 cc/min
* Bilirubin < 2 mg/dL

  * If bilirubin is 2-3 mg/dL, but direct bilirubin is normal then patient will be considered eligible
* Aspartate aminotransferase (AST) < 3 x upper limit of normal
* DONOR: HLA-identical sibling (6/6); the donor must be determined to be an human leukocyte antigen (HLA)-identical sibling (6/6) by serologic typing for class (A, B) and low resolution molecular typing for class II (DRB1)
* DONOR: Matched unrelated donor (10/10); high resolution molecular typing at the following loci is required: HLA-A, -B, -C, -DRB1, and -DQB1
* DONOR: the donor must be healthy and must be an acceptable donor as per institutional standards for stem cell donation
* DONOR: the donor must have no significant cardiopulmonary, renal, endocrine, or hepatic disease
* DONOR: there is no donor age restriction if the donor is a matched sibling
* DONOR: syngeneic donors are not eligible

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Devine, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (21):
- United States (21):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Devine SM, Owzar K, Blum W, Mulkey F, Stone RM, Hsu JW, Champlin RE, Chen YB, Vij R, Slack J, Soiffer RJ, Larson RA, Shea TC, Hars V, Sibley AB, Giralt S, Carter S, Horowitz MM, Linker C, Alyea EP. Phase II Study of Allogeneic Transplantation for Older Patients With Acute Myeloid Leukemia in First Complete Remission Using a Reduced-Intensity Conditioning Regimen: Results From Cancer and Leukemia Group B 100103 (Alliance for Clinical Trials in Oncology)/Blood and Marrow Transplant Clinical Trial Network 0502. J Clin Oncol. 2015 Dec 10;33(35):4167-75. doi: 10.1200/JCO.2015.62.7273. Epub 2015 Nov 2. PMID 26527780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2004 and 2011, 121 participants were registered and received transplants at 21 centers.
Pre-assignment Details: Seven (7) participants were excluded from the all analyses after they were deemed ineligible.
Groups:
- Treatment (Fludarabine, Busulfan, Allogeneic PBSC): PREPARATIVE REGIMEN: Patients receive fludarabine 30 mg/m^2 IV over 30 minutes on days -7 to -3 and busulfan 0.8 mg/kg IV over 2 hours 4 times per day (every 6 hours) on days -4 and -3.
  GVHD PROPHYLAXIS: Patients receive tacrolimus 0.03 mg/kg (suggested starting dose) PO BID on days -2 with taper between days 90-120, and stopping by days 150-180. Patients also receive methotrexate 5 mg/m^2 IV on days 1, 3, 6, and 11 and rabbit antithymocyte globulin 2.5 mg/kg IV over 4-6 hours on days -4 through -2.
  ALLOGENEIC PBSC: Patients undergo allogeneic PBSC transplant on day 0. Patients then receive filgrastim 5 or 10 mcg/kg SC daily beginning on day 12 and continuing until blood counts recover.
Period: Overall Study
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Started | 114
Completed | 114
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Seven (7) participants were excluded from the all analyses after they were deemed ineligible.
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Number analyzed (Participants) | 114
Age, Continuous [Median (Full Range); unit: years] | 65 [60 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 105
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 114
Transplant Donor Type [Number; unit: participants]
  Matched unrelated donor | 59
  Matched related donor | 55

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Disease Free Survival In Unrelated Donor Recipient Group
Description: Percentage of participants who were alive and relapse free at 2 years for patients who were matched with an unrelated donor for transplant. The 2 year disease free survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
  A relapse is defined as any of the following:
  * Reappearance of leukemia blasts cells in peripheral blood
  * >5% blasts in the marrow, not attributable to another cause (e.g., bone marrow regeneration)
  * If there are no circulating blasts, but the marrow contains 5-20% blasts, a repeat bone marrow ≥ 1 week later with >5% blasts is necessary to meet the criteria for relapse
  * The development of extramedullary leukemia or leukemic cells in the cerebral spinal fluid
Time Frame: 2 years
Population: Participants who received a matched unrelated donor were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Number analyzed (Participants) | 59
percentage of participants | 40 [29 to 55]

2. Secondary Outcome: 2 Year DFS for All Patients
Description: Percentage of participants who were alive and relapse free at 2 years for all patients. The 2 year disease free survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Number analyzed (Participants) | 114
percentage of participants | 42 [33 to 52]

3. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Percentage of patients who died due to causes other than relapse
Time Frame: Up to 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Number analyzed (Participants) | 114
percentage of patients | 16

ADVERSE EVENTS:
Arm/Group | Treatment (Fludarabine, Busulfan, Allogeneic PBSC)
Serious Adverse Events (participants affected / at risk) | 38/114
Other Adverse Events (participants affected / at risk) | 109/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Fludarabine, Busulfan, Allogeneic PBSC) (N=114)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (24)
Hemolysis (Blood and lymphatic system disorders) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac pain (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 3 (4)
Vision blurred (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 16 (25)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (4)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 8 (15)
Oral pain (Gastrointestinal disorders) | 1 (3)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 5 (5)
Death NOS (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 10 (12)
Fatigue (General disorders) | 15 (23)
Fever (General disorders) | 7 (7)
General symptom (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Bladder infection (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Infectious colitis (Infections and infestations) | 2 (2)
Lip infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 7 (9)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (6)
Wound infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (12)
Alkaline phosphatase increased (Investigations) | 11 (17)
Aspartate aminotransferase increased (Investigations) | 10 (12)
Blood bilirubin increased (Investigations) | 7 (8)
Creatinine increased (Investigations) | 13 (16)
INR increased (Investigations) | 2 (3)
Laboratory test abnormal (Investigations) | 4 (8)
Leukocyte count decreased (Investigations) | 5 (8)
Lymphocyte count decreased (Investigations) | 6 (13)
Neutrophil count decreased (Investigations) | 21 (26)
Platelet count decreased (Investigations) | 28 (52)
Serum cholesterol increased (Investigations) | 1 (3)
Weight gain (Investigations) | 7 (13)
Weight loss (Investigations) | 7 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 15 (24)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (12)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (12)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 14 (21)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (6)
Serum potassium decreased (Metabolism and nutrition disorders) | 9 (12)
Serum potassium increased (Metabolism and nutrition disorders) | 6 (9)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (8)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 6 (7)
Dysgeusia (Nervous system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (5)
Confusion (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 6 (9)
Insomnia (Psychiatric disorders) | 5 (5)
Psychosis (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 2 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (8)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 20 (31)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (8)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (13)
Hypotension (Vascular disorders) | 11 (15)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Fludarabine, Busulfan, Allogeneic PBSC) (N=114)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 45 (49)
Hemoglobin decreased (Blood and lymphatic system disorders) | 55 (141)
Hemolysis (Blood and lymphatic system disorders) | 4 (6)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (3)
Cardiac disorder (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 3 (4)
Left ventricular failure (Cardiac disorders) | 5 (6)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Ear disorder (Ear and labyrinth disorders) | 2 (5)
Ear pain (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 3 (4)
Hearing impaired (Ear and labyrinth disorders) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 7 (11)
Cataract (Eye disorders) | 5 (6)
Conjunctivitis (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 15 (38)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 6 (6)
Eye pain (Eye disorders) | 2 (2)
Optic nerve disorder (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 4 (4)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (14)
Anal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 26 (35)
Diarrhea (Gastrointestinal disorders) | 52 (80)
Dry mouth (Gastrointestinal disorders) | 18 (35)
Dyspepsia (Gastrointestinal disorders) | 18 (29)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 16 (18)
Enteritis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (8)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 49 (76)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (3)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (30)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 20 (23)
Edema limbs (General disorders) | 23 (35)
Fatigue (General disorders) | 60 (128)
Fever (General disorders) | 27 (31)
Gait abnormal (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Hypothermia (General disorders) | 2 (2)
Ill-defined disorder (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 15 (18)
Hypersensitivity (Immune system disorders) | 9 (9)
Abdominal infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 4 (5)
Catheter related infection (Infections and infestations) | 1 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 3 (4)
Ileal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 11 (13)
Infectious colitis (Infections and infestations) | 1 (1)
Infectious meningitis (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (2)
Opportunistic infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 7 (7)
Scrotal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 11 (14)
Sinusitis (Infections and infestations) | 5 (6)
Skin infection (Infections and infestations) | 6 (7)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (11)
Urinary tract infection (Infections and infestations) | 6 (7)
Vaginal infection (Infections and infestations) | 1 (1)
Viral hepatitis (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
Venous injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 7 (14)
Alanine aminotransferase increased (Investigations) | 41 (87)
Alkaline phosphatase increased (Investigations) | 34 (70)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 45 (106)
Blood bilirubin increased (Investigations) | 23 (34)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 50 (116)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
INR increased (Investigations) | 10 (13)
Laboratory test abnormal (Investigations) | 7 (12)
Leukocyte count decreased (Investigations) | 28 (54)
Lymphocyte count decreased (Investigations) | 26 (44)
Neutrophil count decreased (Investigations) | 95 (157)
Platelet count decreased (Investigations) | 97 (206)
Serum cholesterol increased (Investigations) | 10 (17)
Weight gain (Investigations) | 13 (17)
Weight loss (Investigations) | 12 (16)
Anorexia (Metabolism and nutrition disorders) | 37 (53)
Blood glucose increased (Metabolism and nutrition disorders) | 60 (133)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 8 (8)
Iron overload (Metabolism and nutrition disorders) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 29 (52)
Serum calcium decreased (Metabolism and nutrition disorders) | 26 (48)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (7)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 50 (87)
Serum magnesium increased (Metabolism and nutrition disorders) | 3 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 13 (15)
Serum potassium decreased (Metabolism and nutrition disorders) | 30 (42)
Serum potassium increased (Metabolism and nutrition disorders) | 22 (32)
Serum sodium decreased (Metabolism and nutrition disorders) | 40 (76)
Serum sodium increased (Metabolism and nutrition disorders) | 6 (10)
Serum triglycerides increased (Metabolism and nutrition disorders) | 10 (13)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 13 (23)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (24)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 17 (22)
Dysgeusia (Nervous system disorders) | 9 (18)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 28 (37)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 4 (6)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8)
Seizure (Nervous system disorders) | 2 (3)
Sinus pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (6)
Tremor (Nervous system disorders) | 10 (16)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 11 (14)
Confusion (Psychiatric disorders) | 9 (15)
Depression (Psychiatric disorders) | 12 (24)
Insomnia (Psychiatric disorders) | 19 (30)
Psychosis (Psychiatric disorders) | 1 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 2 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 10 (18)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 3 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (5)
Irregular menstruation (Reproductive system and breast disorders) | 3 (4)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (38)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 (52)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (31)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (27)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (36)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 75 (151)
Skin disorder (Skin and subcutaneous tissue disorders) | 8 (11)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (4)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (3)
Hemorrhage (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 39 (68)
Hypotension (Vascular disorders) | 26 (34)
Thrombosis (Vascular disorders) | 4 (4)
Vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less